CLINICAL TRIAL: NCT01965418
Title: A Clinical Evaluation on Traditional Chinese Medicine Diagnosis and Treatment Program Blocking and Reversing Hepatitis B-related Liver Fibrosis - a Randomized, Controlled, Double-blind, Multi-center Clinical Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013ZX10005002
Record Dates: First submitted 2013-10-16; First posted 2013-10-18 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Liver Fibrosis; Chronic Hepatitis B
MeSH Terms: conditions — Liver Cirrhosis; Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fufang Biejia Ruangan Tablet (Active Comparator): Fufang Biejia Ruangan Tablet will be administered to all of subjects in this arm.
  Interventions: Drug: Fufang Biejia Ruangan Tablet
- placebo (Placebo Comparator): placebo of Fufang Biejia Ruangan Tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fufang Biejia Ruangan Tablet
  Arms: Fufang Biejia Ruangan Tablet
Drug: Placebo
  Arms: placebo

SUMMARY:
This research puts liver biopsy as the enrollment screening criteria and the primary efficacy assessment indicators. Patients at different developmental stages of hepatitis B related liver fibrosis are respectively diagnosed and treated by Traditional Chinese medicine to determine optional diagnosis and treatment plan of traditional Chinese medicine to screen the advantage-treated population and to establish a treatment program, which can save national medical resources, for clinical application of Traditional Chinese medicine Diagnosis and Treatment blocking and reversing hepatitis B-related liver fibrosis. The research can help to build automation pathological analysis and diagnosis systems and non-invasive clinical assessment criteria and models of liver fibrosis which can be applied in clinical. It can also help to realize electronic patient data collection and management, to establish patients management centre and follow-up database. Then it will help to improve clinical efficacy of being blocked and reversed chronic hepatitis B related liver fibrosis by Chinese medicine Diagnosis and Treatment program, to reduce the incidence of liver cirrhosis and hepatitis B-related mortality, to prolong patients' survival and improve patients' quality of life, to make clinical efficacy, which is about Traditional Chinese Medicine blocking and revering chronic hepatitis B-related liver fibrosis, increase by 15% or more .

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria of chronic hepatitis B related liver fibrosis:

1. Age from 18 to 65 years old, male or female;
2. Consistent with the diagnosis criteria of chronic hepatitis B;
3. liver fibrosis(liver biopsy) stage F ≥ 3 (Ishak), HBV DNA ≥ 104 copies / ml (or ≥ 2000 IU / ml) were;
4. TCM syndrome type: blood stasis, blood deficiency with toxic heat retention;
5. Not taking over nucleoside antiviral in one year, no drug treatment of liver fibrosis in six months;
6. Signed informed consent.

Exclusion Criteria:

1. liver fibrosis(Liver biopsy) stage F <3 (Ishak);
2. Combined with other severe chronic hepatitis, cirrhosis, liver cancer and other severe or end-stage liver disease;
3. Accompanied by uncontrollable heart, kidney, lung, endocrine, blood, metabolic and gastrointestinal serious primary disease; or mental illness;
4. Pregnant or lactating women;
5. Patients with allergic constitution or allergic to TCM used;
6. Not be prescribed medication, poor compliance, incomplete data affecting the efficacy and safety of those judgments;
7. Patients unsuitable for this trial in Researchers' consideration;
8. Co-infection with other viral liver disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Liver histological changes | before treatment and after 48 weeks twice

CONTACTS AND LOCATIONS:
Overall Officials: Yongping Yang, Master, Principal Investigator — Beijing 302 Hospital
Locations (1):
- 302 Military Hospital of China, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Rong G, Chen Y, Yu Z, Li Q, Bi J, Tan L, Xiang D, Shang Q, Lei C, Chen L, Hu X, Wang J, Liu H, Lu W, Chen Y, Dong Z, Bai W, Yoshida EM, Mendez-Sanchez N, Hu KQ, Qi X, Yang Y. Synergistic Effect of Biejia-Ruangan on Fibrosis Regression in Patients With Chronic Hepatitis B Treated With Entecavir: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial. J Infect Dis. 2022 Mar 15;225(6):1091-1099. doi: 10.1093/infdis/jiaa266. PMID 32437567
- [Derived] Qu J, Yu Z, Li Q, Chen Y, Xiang D, Tan L, Lei C, Bai W, Li H, Shang Q, Chen L, Hu X, Lu W, Li Z, Chen D, Wang X, Zhang C, Xiao G, Qi X, Chen J, Zhou L, Chen G, Li Y, Zeng Z, Rong G, Dong Z, Chen Y, Lou M, Wang C, Lu Y, Zhang C, Yang Y. Blocking and reversing hepatic fibrosis in patients with chronic hepatitis B treated by traditional Chinese medicine (tablets of biejia ruangan or RGT): study protocol for a randomized controlled trial. Trials. 2014 Nov 10;15:438. doi: 10.1186/1745-6215-15-438. PMID 25381721